CLINICAL TRIAL: NCT05442788
Title: A Phase Ib, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HB0017 Following Multiple Dose in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of HB0017 in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0017-02
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HB0017 150mg (Experimental): 10 subjects is randomly assigned to receive HB0017 150mg or matching placebo at a ratio of 4:1.
  Interventions: Biological: HB0017 150mg or matching placebo
- HB0017 300mg (Experimental): 10 subjects is randomly assigned to receive HB0017 300mg or matching placebo at a ratio of 4:1.
  Interventions: Biological: HB0017 300mg or matching placebo
- HB0017 450mg (Experimental): 10 subjects is randomly assigned to receive HB0017 450mg or matching placebo at a ratio of 4:1.
  Interventions: Biological: HB0017 450mg or matching placebo

INTERVENTIONS:
Biological: HB0017 150mg or matching placebo — Each subject receive injection at week0(Day1), week 3(Day22), week 6(Day43) and week 9(Day64), respectively.
  Arms: HB0017 150mg
Biological: HB0017 300mg or matching placebo — Each subject receive injection at week0(Day1), week 3(Day22), week 6(Day43) and week 9(Day64), respectively.
  Arms: HB0017 300mg
Biological: HB0017 450mg or matching placebo — Each subject receive injection at week0(Day1), week 3(Day22), week 6(Day43) and week 9(Day64), respectively.
  Arms: HB0017 450mg

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation Phase Ib study to evaluate the safety, tolerability, and pharmacokinetics of HB0017 following multiple dose in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, placebo-controlled, multiple dose-escalation study to evaluate the safety, tolerability, PK and immunogenicity of HB0017 in patients with Moderate to severe plaque psoriasis be given HB0017 at doses of 150mg, 300mg and 450mg or placebo by SC administration every 3 weeks. Each cohort of 10 subjects is randomly assigned to receive either a single dose of HB0017 or matching placebo at a ratio of 4:1. Each subject receive injection at week0(Day1), week 3(Day22), week 6(Day43) and week 9(Day64), respectively. After the evaluation and unblinding is completed at week 12(Day 85), the subjects in placebo group completed all study periods, and the HB0017 group continued to be followed up until the end of week 20(D141).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for study entry:

1. Male or female subjects age≥18 and ≤60 years.
2. Weight≥50kg,Body Mass Index(BMI)≥18 and ≤28kg/m2.
3. Subjects with stable moderate to severe chronic plaque psoriasis of ≥6 months' duration with or without psoriatic arthritis.
4. Baseline subjects with moderate or severe plaque psoriasis, defined as below: body surface area (BSA) involvement ≥10%,Psoriasis Area and Severity Index (PASI) ≥12, Static Physician Global Assessment (sPGA) ≥3.
5. Candidates for systemic therapy or phototherapy judged by the investigator or accepted systemic therapy or phototherapy at least one time before.
6. Women who are at childbearing age(not pregnant or breast-feeding), and subjects and their partners voluntarily use contraceptive methods deemed effective by the investigator during treatment and for at least 6 months after the last study medication.
7. During the study, Prolonged exposure to sunlight and the use of ultraviolet health rooms or other ultraviolet light sources must be avoided.
8. Informed consent must be obtained in writing for all subjects enrolled into the study.
9. Subjects must be willing and able to complete study procedures and follow-up examinations.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study entry:

1. Screening for psoriasis other than chronic plaque (such as pustular erythroderma and guttate psoriasis).
2. Drug-induced psoriasis (including, but not limited to, new psoriasis or exacerbations of psoriasis caused by beta blockers calcium channel inhibitors or lithium).
3. Have other active skin diseases or skin infections (bacterial, fungal or viral) that may interfere with clinical evaluation of psoriasis.
4. Patients with symptoms or signs of progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, nerve, mental or brain diseases, or other chronic diseases that are not suitable for the study.
5. Screening of patients with radiographic abnormalities within the preceding 3 months suggesting pulmonary infection or fibrosis or tumor.
6. History of exposure to active tuberculosis (TB); History of TB infection; TB lesions on chest X-ray/chest CT. QuantiFERON®-TB Gold orT-SPOT®.TB positive in the 6 weeks prior to first administration.
7. Having any severe systemic or local infection within 2 months prior to screening.
8. History of chronic recurrent infectious diseases, including but not limited to chronic kidney infections chronic chest infections (such as bronchiectasis) complex urinary tract infections (recurrent pyelonephritis or chronic cystitis) or open,drainage or skin wound infections or ulcers.
9. History of underlying or active granulomatous infection, including histoplasmosis or coccosis.
10. Non-tuberculous mycobacterial infection or opportunistic infection (e.g.,cytomegalovirus infection with pneumocystis carinii and aspergillosis) within 6 months prior to screening.
11. Subjects whose blood pressure is higher than 140 mmHg/90 mmHg (if their blood pressure exceeds this threshold, they may be retested after at least 10 minutes of quiet rest at the discretion of the investigator; if their blood pressure is lower than this threshold, they may be enrolled; Patients who have a history of hypertension but have stable blood pressure control and meet the requirements of the program can be included in the group).
12. Having unstable cardiovascular disease was defined as having had a clinical deterioration in the last 3 months (e.g., unstable angina or rapid atrial fibrillation) or having been hospitalized for heart disease in the last 3 months.
13. Significant abnormalities in heart rate, ECG and respiratory system, and has been judged to be of clinical significance by the investigator.
14. Liver, kidney and blood abnormalities, including:

    1. Glutamate aminotransferase (AST) or aspartate aminotransferase (ALT) exceeds 2 times the normal value (if the first measured value of AST and ALT exceeds this limit, the retest can be carried out once within 7 days; if the retest value is lower than the standard limit, the retest value is acceptable).
    2. Hemoglobin (HGB)< 100g/L.
    3. Platelet count(PLT)<100*109/L.
    4. White blood cells(WBC) <3.5*109/L.
    5. absolute value of neutrophils（NEUT#）<2*109/L.
    6. Serum creatinine was higher than the upper limit of normal value.
    7. Abnormal results of other laboratory tests may, in the investigator's judgment, affect the completion of the test or interfere with the test results.
15. Patients who have had malignant tumors (except basal cell carcinoma of the skin and cervical cancer in situ, which have been cured and have no signs of recurrence) or lymphoproliferative diseases, or cervical diseases caused by HPV.
16. Patients who were allergic to any component of the study drug, or had a history of severe allergic reaction to monoclonal antibodies, or were admitted to the study as determined by the investigator to be at risk of allergy.
17. History of alcohol or drug abuse or have positive results of drug abuse at screening.
18. Hepatitis C virus antibody positive, human immunodeficiency virus positive, treponema pallidum antibody positive;Hepatitis B virus screening program includes hepatitis B virus surface antigen (HbsAg), hepatitis B virus surface antibody (HBsAb) and hepatitis B virus core antibody (HBcAb) : HbsAg positive subjects, screening failure,Only HBcAb positive subjects must be further tested for Hepatitis B virus (HBV) DNA load. If HBV DNA is positive or above the upper limit of normal, screening will fail.
19. Use of topical anti-psoriasis therapy (including topical use of non-weak glucocorticoids, retinoids, vitamin D3 derivatives, salicylic acid, anthracene, etc.) within 2 weeks prior to screening.
20. Use of anti-rheumatism drugs (DMARDs), antimalarial drugs, interferon and lithium within 4 weeks prior to screening.
21. Use of physical therapy (including photochemotherapy, uv therapy, self-therapy on tanning beds, etc.) within 4 weeks prior to screening.
22. Use of systemic nonbiological psoriasis therapy (glucocorticoids, retinoids, ciclosporin , methotrexate, Tripterygium wilfordii, azathioprine, Mycophenolate Mofetil, the treatment of psoriasis related Chinese medicine,etc.) within 4 weeks prior to screening.
23. Participation in another research 3 months prior to screening or now.
24. Have received or plan to receive any live vaccines 2 months prior to screening.
25. Treatment with biological agents(secukinumab, Ixekizumab,or other IL-17 antibodies≤6 months prior to screening.
26. Treatment with Natalizumab, Rituximab, Alemtuzumab, Abatacept,or other drugs that regulate B or T cells) ≤6 months prior to screening.
27. Before screening, the elution period of the following biologics was shorter than the following: Etanercept, Infliximab and Adalimumab < 60 days; Ustekinumab, Risankizumab or other interleukin-23 antagonists < 6 months; Or other anti-psoriasis treatments not listed and within its 5 half-life.
28. Previous or current autoimmune diseases (e.g. Rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome,etc.).
29. Organ transplantation (except corneal transplantation more than 3 months prior to the first administration).
30. History of demyelinating disease (including myelitis) or neurological symptoms suggestive of demyelinating disease, or have a family history of demyelinating disease.
31. History of neurological or mental disorders, such as epilepsy, dementia, poor compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent AE/SAEs | From baseline through week 20
Elimination half-life (T1/2) | From baseline through week 20
Area under drug-time curve (AUC) | From baseline through week 20
Total clearance (CL/F) | From baseline through week 20
Maximum serum concentrations (Cmax) | From baseline through week 20
Mean retention time (MRT) | From baseline through week 20
Volume of distribution (Vz/F) | From baseline through week 20
Peak time(Tmax) | From baseline through week 20

SECONDARY OUTCOMES:
PASI 75 | Week 12
  Proportion of subjects who achieve PASI 75 response or higher at week 12
PASI 90 | Week 12
  Proportion of subjects who achieve PASI 90 response or higher at week 12
PASI 100 | Week 12
  Proportion of subjects who achieve PASI 100 response at week 12
sPGA | Week 12
  Proportion of subjects who achieve sPGA 0 or 1 at week 12
Immunogenicity | From baseline through week 20
  Immunogenicity: number and percentage of subjects with ADA positive anti-HB0017 antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Congjun Jiang, Master, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang C, Du Y, Liu X, Wang J, Ge C, Xu J, Wang S, Li B, Zhu G, Zhang W, Qian Q, Ma C, Zhu X, Zhan Y, Yang Y. Safety, tolerability, pharmacokinetics and efficacy of HB0017, a humanized monoclonal antibody that targets interleukin-17A, in healthy participants and patients with moderate-to-severe plaque psoriasis. Br J Dermatol. 2023 Dec 20;190(1):28-36. doi: 10.1093/bjd/ljad315. PMID 37669307